CLINICAL TRIAL: NCT04225819
Title: Adjunctive Treatment With Vitamin D3 in Patients With Active IBD (ACTIVATED): A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Adjunctive Treatment With Vitamin D3 in Patients With Active IBD
Acronym: ACTIVATED
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol is being modified.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ashwin Ananthakrishnan, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P003843
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: IBD; Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis; Vitamin D3 Deficiency
Keywords: Vitamin D3; Cholecalciferol; IBD; Inflammatory Bowel Disease; Adjunctive treatment; Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 supplement (Experimental): Two- 5,000 IU capsules, taken daily with a meal
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Two placebo capsules, taken daily with a meal
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Softgel capsules containing 5,000 IU cholecalciferol (Vitamin D3), sunflower oil, beef gelatin, glycerin, water
  Other Names: cholecalciferol
  Arms: Vitamin D3 supplement
Other: Placebo — Sfotgel capsules containing sunflower oil, beef gelatin, glycerin, water
  Arms: Placebo

SUMMARY:
Inflammatory bowel disease ((IBD), which includes Crohn's disease (CD) and ulcerative colitis (UC)), is a chronic, immune-mediated disease characterized by recurrent episodes of relapse. The incidence of IBD is increasing worldwide and poses as a burden that reduces quality of life and has a significant impact on health care resources.

The advent of monoclonal antibodies to tumor necrosis factor-α (anti-TNF) has revolutionized treatment of IBD, improving rates of remission and reducing hospitalizations and surgeries. Nevertheless, many patients do not adequately respond to these therapies or lose response over time. Thus, there is an important need for novel immunomodulating agents to improve our ability to achieve remission.

Besides its traditional role in bone homeostasis, several studies have recognized the important role Vitamin D plays in modulating the immune response, cancer, and cardiovascular disease. Specifically, Vitamin D may mediate immunity by modulating autophagy in leukocytes and regulating the gut microbiome. Thus, Vitamin D may play an important role in IBD. Furthermore, evidence suggests that the effect of vitamin D may be mediated through the TNF-α pathway, suggesting a synergy with anti-TNF therapy.

This is a randomized, double blind, placebo-controlled trial to study the effect of Vitamin D3 as an adjunct therapy for patients with active CD, UC, or IBD unspecified who are undergoing anti-TNF induction therapy.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of CD, UC, or IBD-unspecified
* Initiating anti-TNF therapy for IBD within 2 weeks of baseline/randomization
* Other non-anti-TNF IBD medications must remain stable during the treatment period with the exception of tapering of corticosteroids.
* Recent (within 6 months) objective evidence of active IBD on colonoscopy along with elevated inflammatory markers (C-reactive protein >8 mg/L or fecal calprotectin >150 mcg/g)
* Current disease activity defined as a Harvey Bradshaw index > 4 at baseline (week 0) for CD subjects or Simple Clinical Colitis Activity Index > 2 at baseline (week 0) for UC subjects.
* Fecal Calprotectin level >150 mcg/g

Exclusion Criteria:

* Inability to provide informed consent or unwilling or unlikely to comply with the requirements of the study.
* Female subjects who are pregnant, lactating, or intending to become pregnant during the study period
* Known intolerance or hypersensitivity to oral vitamin D3 supplementation
* Plasma 25(OH)D > 60 ng/mL
* Known celiac disease or subjects with a positive screen for celiac disease (elevated tissue transglutaminase antibodies)
* Serum calcium >11 mg/dL
* History of hyperparathyroidism
* History of renal calculi or chronic kidney disease
* Initiation of anti-TNF treatment for extra-intestinal symptoms alone
* Evidence of untreated infection (e.g. Clostridium difficile)
* History of chronic pancreatitis
* History of cystic fibrosis
* History of gastric bypass
* Presence of stoma or J-pouch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) outcome | 14 weeks
  Patients will complete the SIBDQ questionnaire to measure disease activity at baseline, week 6 and week 14.
stool microbiome in IBD patients | 14 weeks
  Stool samples will be taken at baseline and week 14 to assess change in stool microbiome
serum cathelicidin levels | 14 weeks
  Serum samples will be taken at baseline and week 14 to measure serum cathelicidin levels
HBI | 14 weeks
  Patients with Crohn's Disease will complete the Harvey Bradshaw Index questionnaire to measure disease activity at baseline, week 6 and week 14
SCCAI | 14 weeks
  Patients with Ulcerative Colitis will complete the Simple Clinical Colitis Activity Index questionnaire to measure disease activity at baseline, week 6 and week 14

SECONDARY OUTCOMES:
fecal calprotectin | 14 weeks
  Stool samples will be taken at baseline and week 14 to assess change in fecal calprotectin levels
plasma 25(OH)D levels. | 14 weeks
  Plasma samples will be taken at baseline and week 14 to measure 25(OH)D levels

CONTACTS AND LOCATIONS:
Overall Officials: Ashwin Ananthakrishnan, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No